CLINICAL TRIAL: NCT04037449
Title: Prospective Randomized Study to Measure the Effect of Bilateral Transversus Abdominis Plane (TAP) Block in the Analgesic Control of Patients With Acute Pancreatitis (AP) and Uncontrolled Pain
Brief Title: Transversus Abdominis Plane Block in the Analgesia of Acute Pancreatitis
Acronym: TAPA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Consorci Sanitari Integral (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19/35
Record Dates: First submitted 2019-05-27; First posted 2019-07-30 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Pancreatitis, Acute
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP block (Experimental): Transversus Abdominis Plane (TAP) block technique will be carried out by a restricted group of anaesthesiologists. Standard monitoring will be applied to all patients, which will include pulse oximetry, electrocardiogram and non-invasive monitoring of blood pressure.
  Interventions: Procedure: TAP block
- Conventional analgesia (Active Comparator): Patients be given conventional endovenous analgesia, and morphine 2 mg / ev every 15 minutes until the level of pain measured by a Visual Analogue Scale (VAS) ≤ 3
  Interventions: Other: Conventional analgesia

INTERVENTIONS:
Procedure: TAP block — With the patient placed in the supine position, after asepsis of the skin with chlorhexidine, bilateral TAP blockage will be carried out under ultrasound control. We will use a high frequency linear transducer (12-15 MHz) on one side of the abdominal wall, at the level of the mid-axillary line, between the costal margin and the iliac crest. At this level we can identify three muscle layers, from superficial to deep: external oblique muscle, internal oblique muscle and transverse muscle of the abdomen. We will move the transducer more laterally to locate the most posterior border of the internal oblique and transverse muscles. It is at this level that we perform the posterior TAP blockade: we administer 10 ml of 2% Mepivacaine plus 10 ml of 0.5% Bupivacaine between the fasciae of the internal oblique muscle and the transverse muscle of the abdomen and observe an appropriate diffusion pattern of local anesthetics
  Arms: TAP block
Other: Conventional analgesia — Intravenous dexketoprofen 50 mg / 8 hours, alternate with intravenous paracetamol 1g / 8 hours. If allergy to Nonsteroidal anti-inflammatory drugs (NSAIDs) or in case of renal failure: Intravenous metamizol 2g / 8 hours alternate with intravenous paracetamol 1g / 8 hours.
  Rescue Analgesia: intravenous morphine (2 mg every 15 minutes until VAS less or equal to 3)
  Arms: Conventional analgesia

SUMMARY:
Background Severe abdominal pain is a hallmark of acute pancreatitis (AP). A control pain is often difficult. Transversus Abdominis Plane (TAP) block has been used in pain control in patients with exacerbation of chronic pancreatitis.

Objectives To evaluate the effect of Bilateral Blockade of the Abdominal Transverse Muscle Plane (TAP Block) in the analgesic control of patients with acute pancreatitis; compared to standard intravenous analgesia.

Methods A randomized controlled trial of parallel groups will be conducted. The Study will have a multicenter development. Study population: Adult patients admitted for episode of AP, with uncontrolled pain (visual analogue scale (VAS) equal to or greater than 5 after the administration of standard analgesia. Randomization Groups: Group A: Patients who will undergo TAP block as analgesic procedure added to standard analgesia. Group B: Patients to whom morphine 2 mg / ev will be administered as analgesic procedure added to standard analgesia.

Timing of pain determination (Visual Analogue Scale, VAS):

* Before conventional analgesia
* Immediately before Randomization
* 15 minutes after the administration of the analgesic treatment object of the study.
* One hour after the procedure.
* Every 8 hours, during the next 4 days or until discharge of the patient.
* Whenever the patient needs a dose of supplemental rescue analgesia. Analysis of data All results will be evaluated according to the initial "intention to treat". There will be a blinded assessment of the results after the last patient in the trial has completed the follow-up. The results will be presented as relative risks with their corresponding confidence intervals. P <0.05 will be considered statistically significant. In case of imbalance between the two treatment groups, a multivariate logistic regression is used to correct possible confounding factors.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute pancreatitis according to modified Atlanta criteria .
* Patients with the ability to understand the VAS scale and express their level of pain.
* Patients over 18 years old.
* Uncontrolled pain, with VAS ≥ 5 after the administration of standard analgesia.
* Material and technical possibility of performing the TAP technique immediately after randomization.
* Informed consent of the participating patients for inclusion in the study.
* Informed consent of the participating patients for the administration of TAP.
* Normality of coagulation levels

Exclusion Criteria:

* Patients with American Society of Anaesthesia (ASA) levels IV and V
* Patients with chronic pancreatitis
* Pregnancy
* Patients with chronic treatment with morphic medication

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2020-11-30 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Change of pain levels (VAS) after the intervention | Baseline (Before the intervention), 15 minutes after the intervention, 1 hour after the intervention, 8 hours after the intervention, 16 hours after the intervention, 24 hours after the intervention
  To assess the VAS value in order to measure the time elapsed from the intervention until reaching the appropriate level of analgesic efficacy. Analgesic efficacy is defined as the patient having a pain VAS value ≤ 3.

SECONDARY OUTCOMES:
Complications | through study completion, an average of 30 days
  Complications related to the analgesic technique used, either by the administration procedure or as a side effect

IPD SHARING:
Plan to Share IPD: No